CLINICAL TRIAL: NCT06333327
Title: Multielectrode Radiofrequency Balloon for Atrial Fibrillation Catheter Ablation: A Multicenter Real-World Experience
Brief Title: Multicenter Registry of Atrial Fibrillation Ablation With Radiofrequency Balloon Catheter
Acronym: COLLABORATE
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, MD, PhD, Universitair Ziekenhuis Brussel
Other Study IDs: 1432022000278
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: Radiofrequency, Ablation, Single-shot
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pulmonary vein isolation with the multielectrode radiofrequency balloon catheter — Pulmonary vein isolation with the multielectrode radiofrequency balloon catheter

SUMMARY:
All consecutive patients with paroxysmal or persistent atrial fibrillation undergoing pulmonary vein isolation with the radiofrequency balloon catheter (RFB) "Heliostar" (Biosense Webster) will be included in a multicenter observational registry. The aim of the study is to assess the safety and arrhythmic outcome of atrial fibrillation ablation with the RFB in a real-world setting.

DETAILED DESCRIPTION:
All consecutive atrial fibrillation patients undergoing pulmonary vein isolation (PVI) with the novel radiofrequency balloon catheter (RFB) "Heliostar" (Biosense Webster) will be prospectively included in a multicenter observational registry.

PVI with the RFB will be performed as previously described. Briefly, after optimal RFB positioning, confirmed through the correct alignment between the RFB and the pulmonary vein and sufficient electrode-tissue contact, ablation is performed in temperature-controlled mode with unipolar radiofrequency energy. Typically, >2 posterior electrodes are identified on the RFB. The power setting is 15 W and the target electrode temperature is 55° C. The same energy is simultaneously delivered to all electrodes, with a duration of 15-20 s for the posterior and 45-60 s for the non-posterior electrodes. During ablation, pulmonary vein potentials are monitored on the circular diagnostic catheter to evaluate real-time isolation. In the case of pulmonary vein acute reconnection, additional applications are delivered to achieve durable PVI. An esophageal temperature probe will be used to monitor any increase in esophageal temperature.

Follow-up will be performed according to each standard institutional protocol.

Safety endpoints include any major periprocedural complications [e.g. death, atrioesophageal fistula, stroke/transient ischaemic attack, pericardial effusion/tamponade with/without surgical treatment, myocardial infarction, and persistent phrenic palsy] occurring within 7 days post-procedure (except for atrioesophageal fistula). Minor complications will also be reported, including vascular access complications requiring treatment, pericarditis, and transient phrenic palsy.

Efficacy outcome is defined as arrhythmia-free survival during the follow-up. Arrhythmia recurrence is defined as any atrial tachyarrhythmias ≥30 s after a 90-day post-ablation blanking period.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic atrial fibrillation with indication to catheter ablation

Exclusion Criteria:

* age <18 years old
* pregnancy
* any contraindications to catheter ablation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with symptomatic paroxysmal or persistent atrial fibrillation undergoing a first-time pulmonary vein isolation with the multielectrode radiofrequency balloon catheter (HELIOSTAR, Biosense Webster, CA, USA) will be prospectively included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Atrial arrhythmia recurrence after ablation | After 3 months post-ablation.
  The primary outcome endpoint is defined as arrhythmia-free survival during the follow-up. Arrhythmia recurrence is defined as any atrial tachyarrhythmias ≥30 s after a 90-day post-ablation blanking period.
Procedural safety | Up to 7 days post-procedure (except for atrioesophageal fistula or pulmonary vein stenosis)
  The primary safety endpoint included any major periprocedural complications [e.g. death, atrioesophageal fistula, stroke/transient ischaemic attack (TIA), pericardial effusion/tamponade with/without surgical treatment, myocardial infarction, and persistent phrenic palsy] occurring within 7 days post-procedure (except for atrioesophageal fistula). Minor complications, including vascular access complications requiring treatment, pericarditis, and transient phrenic palsy will also be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel Heart Rhythm Management Center, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided